CLINICAL TRIAL: NCT00002578
Title: Phase II Evaluation of Gallium Nitrate (NSC 15200) in Non-Hodgkin's Lymphoma in Patients With Acquired Immunodeficiency Syndrome
Brief Title: Gallium Nitrate in Treating Patients With AIDS-Related Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: DS 96-26; RPCI-DS-96-26; UTHSC-9235011358; NCI-T94-0043D
Record Dates: First submitted 1999-11-01; First posted 2004-05-20 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Lymphoma
Keywords: AIDS-related peripheral/systemic lymphoma; AIDS-related diffuse large cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related small noncleaved cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related lymphoblastic lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Cytarabine; gallium nitrate; Leucovorin; Methotrexate

INTERVENTIONS:
Drug: cytarabine
Drug: gallium nitrate
Drug: leucovorin calcium
Drug: methotrexate

SUMMARY:
RATIONALE: Chemotherapy uses different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of gallium nitrate in treating patients with AIDS-related non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and duration of response in patients with AIDS-related non-Hodgkin's lymphoma treated with gallium nitrate after failure on first-line chemotherapy regimen. II. Determine the qualitative and quantitative toxic effects of this regimen in these patients. III. Determine the pharmacokinetic parameters of this regimen in these patients, and determine if there is a correlation between those parameters and response.

OUTLINE: Patients receive gallium nitrate IV continuously on days 1-7. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients who achieve complete remission (CR) receive 2 additional courses past CR. Patients who relapse after achieving CR may be retreated in the absence of disease progression. Treatment for relapse after a second CR is at the discretion of the principal investigator. Patients with leptomeningeal disease at study entry must receive intrathecal (IT) methotrexate with IV leucovorin calcium or IT cytarabine. Patients who develop leptomeningeal disease while on study may continue treatment with gallium nitrate but must also receive IT methotrexate and leucovorin calcium (with or without radiotherapy) or IT cytarabine. Patients are followed for survival.

PROJECTED ACCRUAL: A total of 20-35 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage I-IV AIDS-related non-Hodgkin's lymphoma Intermediate- or high-grade disease HIV infection documented by ELISA and confirmed by Western blot Must have received at least 1 potentially curative chemotherapy regimen for lymphoma Must be past the hematologic nadir resulting from prior chemotherapy (generally 2 weeks from onset of prior therapy regardless of filgrastim (G-CSF) use) Waiting period waived at the discretion of the principal investigator if patient well-being would be compromised At least 1 site of bidimensionally measurable or evaluable disease (e.g., bone marrow involvement only) History of leptomeningeal disease associated with systemic lymphoma allowed No primary CNS non-Hodgkin's lymphoma A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: At least 6 weeks Hematopoietic: Granulocyte count at least 750/mm3* Platelet count at least 50,000/mm3* Hemoglobin at least 7.5 g/dL* * Unless bone marrow infiltrated by lymphoma Hepatic: Bilirubin less than 1.25 times upper limit of normal AST no greater than 3.0 times normal Renal: Creatinine clearance greater than 60 mL/min Cardiovascular: No myocardial infarction within the past 6 months No history of congestive heart failure No angina No serious arrhythmia requiring treatment Other: No other prior or concurrent malignancy except: Inactive, nonvisceral Kaposi's sarcoma not requiring chemotherapy Curatively treated basal cell or squamous cell skin cancer Curatively treated carcinoma in situ of the cervix No severe, acute opportunistic infection No acute or intermittent infection (other than oropharyngeal candidiasis) requiring treatment within 2 weeks before study entry Not pregnant Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Prior biologic therapy allowed Chemotherapy: See Disease Characteristics No concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy Radiotherapy: Prior radiotherapy allowed No concurrent radiotherapy Surgery: Not specified Other: No concurrent investigational anticancer or anti-infective therapy No concurrent aminoglycosides, amphotericin B, or foscarnet Concurrent required supportive care allowed, including: Non-investigational antiretroviral and antiviral medications Medications for Mycobacterium avium DISEASE CHARACTERISTICS: Histologically proven stage I-IV AIDS-related non-Hodgkin's lymphoma Intermediate- or high-grade disease HIV infection documented by ELISA and confirmed by Western blot Must have received at least 1 potentially curative chemotherapy regimen for lymphoma Must be past the hematologic nadir resulting from prior chemotherapy (generally 2 weeks from onset of prior therapy regardless of filgrastim (G-CSF) use) Waiting period waived at the discretion of the principal investigator if patient well-being would be compromised At least 1 site of bidimensionally measurable or evaluable disease (e.g., bone marrow involvement only) History of leptomeningeal disease associated with systemic lymphoma allowed No primary CNS non-Hodgkin's lymphoma A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: At least 6 weeks Hematopoietic: Granulocyte count at least 750/mm3* Platelet count at least 50,000/mm3* Hemoglobin at least 7.5 g/dL* * Unless bone marrow infiltrated by lymphoma Hepatic: Bilirubin less than 1.25 times upper limit of normal AST no greater than 3.0 times normal Renal: Creatinine clearance greater than 60 mL/min Cardiovascular: No myocardial infarction within the past 6 months No history of congestive heart failure No angina No serious arrhythmia requiring treatment Other: No other prior or concurrent malignancy except: Inactive, nonvisceral Kaposi's sarcoma not requiring chemotherapy Curatively treated basal cell or squamous cell skin cancer Curatively treated carcinoma in situ of the cervix No severe, acute opportunistic infection No acute or intermittent infection (other than oropharyngeal candidiasis) requiring treatment within 2 weeks before study entry Not pregnant Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Prior biologic therapy allowed Chemotherapy: See Disease Characteristics No concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy Radiotherapy: Prior radiotherapy allowed No concurrent radiotherapy Surgery: Not specified Other: No concurrent investigational anticancer or anti-infective therapy No concurrent aminoglycosides, amphotericin B, or foscarnet Concurrent required supportive care allowed, including: Non-investigational antiretroviral and antiviral medications Medications for Mycobacterium avium intracellulare infection Medications for cytomegalovirus (CMV) infection or CMV infection prophylaxis infection Medications for cytomegalovirus (CMV) infection or CMV infection prophylaxis

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 1994-08; Primary Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence P. Leichman, MD, Study Chair — Albany Medical College
Locations (3):
- United States (3):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Roswell Park Cancer Institute, Buffalo, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York